CLINICAL TRIAL: NCT02810470
Title: Acceptability Study of Nutritional Supplements in Hospitalized Elderly Patients Aged for More Than 65 Years
Brief Title: Acceptability Study of Nutritional Supplements in Hospitalized Elderly Patients
Acronym: CNO Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: VAN WYMELBEKE NUTRICIA 2015
Record Dates: First submitted 2016-06-14; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2015-05

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

ARMS (2):
- Cream appreciation tests (Experimental)
  Interventions: Dietary Supplement: Fortimel Compact Protein; Dietary Supplement: Fortimel Cream
- Beverages appreciation tests (Experimental)
  Interventions: Dietary Supplement: Fortimel Compact Protein; Dietary Supplement: Fortimel Cream

INTERVENTIONS:
Dietary Supplement: Fortimel Compact Protein — Each product will be tested by all patients spread over 2 days. A first half of volunteers will start the testing process with the beverages at day 1 and continue with the creams at day 2. The second half of volunteers will process inversely (day 1 = creams, day 2 = beverages). The test order of flavors will be randomly allocated to the volunteers among the list of all possible combinations.
Dietary Supplement: Fortimel Cream — Each product will be tested by all patients spread over 2 days. A first half of volunteers will start the testing process with the beverages at day 1 and continue with the creams at day 2. The second half of volunteers will process inversely (day 1 = creams, day 2 = beverages). The test order of flavors will be randomly allocated to the volunteers among the list of all possible combinations.

SUMMARY:
Malnutrition is a major health problem with serious consequences for the quality of life of elderly people: it increases the number of hospitalizations and lengths of stay, worsens functional dependency and increases morbidity and mortality rates There are numerous recommendations and tools to detect or to manage malnutrition and the prescription of Oral Nutritional Supplements (ONS) can be a solution. As the elderly suffer from food monotony, as well as age-related changes, which may or may not be associated with the presence of disease, it is necessary to ensure full ingestion of the prescribed supplements to optimize the benefits provided by these products. To achieve this it is necessary to know the chemosensory characteristics of foods enjoyed by hospitalized elderly people who are malnourished or at risk of malnutrition. The investigators make the hypothesis that by further optimizing taste and energy content of foods, consumption by the elderly and the health benefits would be improved.

ELIGIBILITY:
Inclusion Criteria:

* Person who have given their written informed consent
* Person aged more than 65 years
* Person cognitively able to participate in tests and to answer questionnaires (Mini Mental Statement Estimation score (MMSE) equal to or greater than 21)
* Person with an Mini Nutritional Status score (MNA) lower than 23.5/30 for risk of malnutrition or malnourished
* Person without known unstable cardiac disease
* Person without high blood pressure

Exclusion Criteria:

* Person who are not covered by national health insurance
* Person suffering from severe illness during the test
* Person with a life expectancy lower than 6 months or with a cancer
* Every person with proven anosmia (total loss of olfaction) from birth or due to physical trauma (head trauma) or disease (acute rhinitis)
* Person with allergy (soya milk) or severe aversion to one of the foods that will be used during the study
* Person with swallowing disorders
* Person with a prescribed strict food diet
* Person with an instable diabetes

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Acceptability of the different tested Oral Nutrition Supplement with different flavors | Hedonic scale after testing at day 2